CLINICAL TRIAL: NCT02310399
Title: Auditory Brainstem Implant (ABI) in Children With No Cochleae or Auditory Nerves
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S14-01010
Record Dates: First submitted 2014-11-28; First posted 2014-12-08 (Estimated); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Hearing Loss, Bilateral (Causes Other Than Tumors)
Keywords: Auditory Brainstem Implant; Deafness; Hearing Loss; ABI
MeSH Terms: conditions — Hearing Loss; Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Pre-lingual Deafness (Experimental): Surgical implantation of the Nucleus ABI541 Auditory Brainstem Implant in prelingiustically deaf children ages 18 months - 5 years
  Interventions: Device: Nucleus ABI541 Auditory Brainstem Implant
- Post-Lingual Deafness (Experimental): Surgical implantation of the Nucleus ABI541 Auditory Brainstem Implant in postlinguistically deaf children < 21 years of age
  Interventions: Device: Nucleus ABI541 Auditory Brainstem Implant

INTERVENTIONS:
Device: Nucleus ABI541 Auditory Brainstem Implant — Surgical implantation of the Nucleus ABI541 Auditory Brainstem Implant device

SUMMARY:
This study is a feasibility study of the Nucleus 24 ABI in children without NF2. It will be conducted as a repeated-measures, single subject experiment in order to accommodate the known variability in cochlear implant clinical results. Data obtained in the course of this study will be compared with the existing published outcome data from children with normal hearing and with cochlear implants (CIs). These comparisons may provide additional useful information about the progress of ABI subjects' performance over time. Also, this may allow the results of the current study to be utilized to design future pivotal studies of the device in the pediatric population.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the clinical safety and efficacy of the Nucleus™ 24 Auditory Brainstem Implant (ABI) in pediatric patients who do not have Neurofibromatosis Type 2 (NF2); specifically, children with total hearing loss due to severe cochlear anomalies, cochlear nerve disorders or failed cochlear implantation. These conditions can include: developmental or acquired cochlear nerve deficiency (CND), cochlear aplasia, post-meningitis cochlear ossification, or cochlear malformation. This study proposes to implant up to 10 pre-linguistic young children (18 mos to 5 yrs. of age) and up to 10 post-linguistic children (<21 yrs of age) with the Nucleus 24 Multichannel ABI in an attempt to demonstrate safety of the surgical procedure and device stimulation and the potential for auditory benefit beyond that experienced with a CI. These children would not qualify for the Nucleus ABI device, as their etiology is not an approved indication such as neurofibromatosis Type 2(NF2). Further, these children do not benefit from conventional hearing aids or cochlear implants.

Two groups of children will be included: Group 1 will include prelingiustic deaf children ages 18 months - 5 years and Group 2 will include postlinguistic deaf children < 21 years of age. Post-operative evaluations will be conducted at the initial activation and at 1, 3, 6, 12, 18, 24, 30, and 36-month intervals post-activation in order to demonstrate the emergence of open-set speech perception abilities prior to study cessation. Experience in the CI literature has shown that a minimum of 2 years of device usage is required for children with pre-lingual hearing impairment to develop some open-set speech perception abilities. While Group 2 is post-linguistic and some may have had significant hearing prior to becoming deaf, the same time intervals will be used for consistency. Blinding or masking procedures are not included in the design, as the presence/absence of a brainstem implant cannot be easily concealed from the device recipients and/or clinical investigators.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Prelinguistic hearing loss (birth-5 years; age at implantation of ABI 18 months-5 years)

• Pre-linguistic hearing loss (birth-5 yrs.; age at ABI 18 months-5yrs) with both:

* MRI +/- CT evidence of one of the following:

  * Cochlear nerve deficiency
  * Cochlear aplasia or severe hypoplasia
  * Severe inner ear malformation
  * Post-meningitis ossification
* When a cochlea is present or patent, lack of significant benefit from CI despite consistent use (>6 mo.)

  * No or limited speech perception ability (limited to pattern perception on closed set testing materials using the CI)
  * Lack of progress in auditory skills development

Group 2: Post-linguistic hearing loss (<21 yrs. of age)

* Post-linguistic hearing loss (<21 yrs. of age) with:

  * Loss or lack of benefit from appropriate CI without the possibility for revision or contralateral implantation. Examples might include:

    * Post-meningitis ossification
    * Bilateral temporal bone fractures with cochlear nerve avulsion
    * Failed revision CI without benefit
  * Previously developed open set speech perception and auditory-oral language skills
* No medical contraindications
* Willing to receive the appropriate meningitis vaccinations
* No or limited cognitive/developmental delays.
* Strong family support
* Reasonable expectations from parents/guardians including a thorough understanding:

  * of potential benefits and limitations of ABI
  * of parental role in rehabilitation
  * that the child may not develop spoken language as a primary communication mode or even sufficient spoken language to make significant academic progress in an aural/oral environment
* Involvement in a rehabilitation program that emphasizes development of auditory skills with or without the use of supplementary visual communication.
* Able to comply with study requirements including travel to investigation sites.
* Informed consent for the procedure from the child's parents/legal guardian.

Exclusion Criteria:

For both Groups 1 and 2:

* Pre- or post-linguistic child currently making significant progress with CI Even for the very young children (18 months of age with 6 months of use), nearly all children with a good auditory signal from their CI will show evidence of improvement in these metrics over time.
* MRI evidence of one of the following:

  * normal cochlea and cochlear nerves or NF2
  * brainstem or cortical anomaly that makes implantation unfeasible
* Clear surgical reason for poor CI performance that can be remediated with revision CI or contralateral surgery rather than ABI.
* Intractable seizures or progressive, deteriorating neurological disorder
* Patients with evidence of Chiari malformation, hydrocephalus, spina bifid a
* Patients with any foreseeable need for a future MRI scan
* Unable to participate in behavioral testing and mapping with their CI. If this appears to be an age effect, ABI will be delayed until we can be assured that the child will be able to participate, as reliable objective measures of mapping are currently not available for mapping these devices.
* Unable to tolerate general anesthesia (cardiac, pulmonary, bleeding diathesis, etc.).
* Need for brainstem irradiation
* Unrealistic expectations on the part of the subject/family regarding the possible benefits, risks and limitations inherent to the procedure and ABI device.
* Unwilling to sign the informed consent.
* Unwilling to make necessary follow-up appointments.

Ages: 18 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
ABI Device Complications | 5 Years from date of surgery
  Study participants will be monitored on a case-by-case basis for ongoing or unanticipated medical complications. Adverse events will be tracked on a case-by-case basis and recorded at the time of occurrence and followed up at resolution. Any adverse events will be reported to the NYUSOM IRB. Should there be concern for the safety of the subjects because of their participation in the study by the investigators or the IRB, the study would be halted at least temporarily and a detailed discussion with the investigators and the IRB would be undertaken.

SECONDARY OUTCOMES:
Audiologic Performance with ABI (Hearing, Speech and Language Assessments) | 36 months from date of surgery
  The following audiometry and speech perception tests will be administered as age-appropriate:
  * Detection audiogram, aided and unaided individual ears
  * IT-MAIS or MAIS
  * LING 6 sound test
  * ESP Low Verbal or Standard- MLV @ 50dB HL
  * PB-k words and phonemes- MLV @ 50dB HL
  * MLNT- recorded @ 60dB SPL
  * LNT- recorded @ 60dB SPL
  * HINT-C- 2 lists of 10 @ 60dB SPL
  * CNC- 50 words @ 60dB SPL
  Each child will receive speech/language intervention using the Comprehensive Assessment of Spoken Language (CASL, Elizabeth Carrow-Woolfolk, 1999) The following tests will be administered when appropriate:
  * The Oral and Written Language Scales (OWLS)
  * Goldman-Fristoe Test of Articulation
  * The Peabody Picture Vocabulary Test (PPVT)
  * The Rossetti Infant-Toddler Language Scale
  * Pre-School Language Scale, (PLS-5)
  * The Expressive Vocabulary Test, 2nd Ed
  * The Peabody Picture Vocabulary Test, 4th Ed

CONTACTS AND LOCATIONS:
Overall Officials: John T. Roland, Jr., MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Cochlear Implant Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Colletti V, Shannon R, Carner M, Veronese S, Colletti L. Outcomes in nontumor adults fitted with the auditory brainstem implant: 10 years' experience. Otol Neurotol. 2009 Aug;30(5):614-8. doi: 10.1097/MAO.0b013e3181a864f2. PMID 19546832
- [Background] Colletti L, Zoccante L. Nonverbal cognitive abilities and auditory performance in children fitted with auditory brainstem implants: preliminary report. Laryngoscope. 2008 Aug;118(8):1443-8. doi: 10.1097/MLG.0b013e318173a011. PMID 18496153
- [Background] Sennaroglu L, Ziyal I, Atas A, Sennaroglu G, Yucel E, Sevinc S, Ekin MC, Sarac S, Atay G, Ozgen B, Ozcan OE, Belgin E, Colletti V, Turan E. Preliminary results of auditory brainstem implantation in prelingually deaf children with inner ear malformations including severe stenosis of the cochlear aperture and aplasia of the cochlear nerve. Otol Neurotol. 2009 Sep;30(6):708-15. doi: 10.1097/MAO.0b013e3181b07d41. PMID 19704357
- [Background] Sennaroglu L, Ziyal I. Auditory brainstem implantation. Auris Nasus Larynx. 2012 Oct;39(5):439-50. doi: 10.1016/j.anl.2011.10.013. Epub 2011 Dec 22. PMID 22196501
- [Background] Colletti L, Shannon RV, Colletti V. The development of auditory perception in children after auditory brainstem implantation. Audiol Neurootol. 2014;19(6):386-94. doi: 10.1159/000363684. Epub 2014 Nov 4. PMID 25377987
- [Background] Colletti L, Wilkinson EP, Colletti V. Auditory brainstem implantation after unsuccessful cochlear implantation of children with clinical diagnosis of cochlear nerve deficiency. Ann Otol Rhinol Laryngol. 2013 Oct;122(10):605-12. PMID 24294682
- See also: NYU Cochlear Implant Center homepage — http://cochlear.med.nyu.edu/